CLINICAL TRIAL: NCT00561132
Title: Effect of Vanadium on Insulin Sensitivity in Patients With Impaired Glucose Tolerance
Brief Title: Study of Vanadium Supplement in Patients With Impaired Glucose Tolerance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Unidad de Investigacion Medica en Epidemiologia Clinica (Other)
Collaborators: Fondo para el Fomento a la Investigacion Medica (Unknown); Doctorado en Farmacologia de la Universidad de Guadalajara (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002/252/129; 173/03/13; FP-2003/073
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Prediabetic State
Keywords: vanadium; insulin sensitivity; impaired glucose tolerance; triglycerides
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Glucose Intolerance | interventions — vanadyl sulfate; Magnesium Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: Vanadyl sulfate
- 2 (Placebo Comparator)
  Interventions: Other: Magnesium oxide

INTERVENTIONS:
Dietary Supplement: Vanadyl sulfate — 50 mg twice daily orally for a period of 4 weeks
  Other Names: Vanadyl sulphate; Vanadyl sulfate hydrate; Vanadyl sulphate hydrate
  Arms: 1
Other: Magnesium oxide — Validation of similar appearance and weight to the intervention component orally 1 unit (<50 mg) twice daily for a period of 4 weeks
  Other Names: Calcinated magnesia; Calcined Magnesite; Magnesia
  Arms: 2

SUMMARY:
The purpose of this study was to evaluate if the vanadium can improve the insulin sensitivity in patients with impaired glucose tolerance. Secondary purpose of this study was to assess changes on metabolic profile, weight and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of impaired glucose tolerance
* Body mass index from 25 to 35 kg/m2
* History of type 2 diabetes mellitus in the first branch

Exclusion Criteria:

* Taking medication with known effects on carbohydrate or insulin metabolism
* Thyroid diseases
* Hepatic diseases

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2003-11; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Changes on insulin sensitivity assessed with a euglycemic-hyperinsulinemic clamp technique | 4 weeks

SECONDARY OUTCOMES:
Changes on metabolic profile | 4 weeks
Changes on anthropometrical measures | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Omar Jacques-Camarena, MD, MSc, Principal Investigator — Unidad de Investigacion Medica en Epidemiologia Clinica; Manuel González-Ortiz, MD, MSc, PhD, Principal Investigator — Unidad de Investigacion Medica en Epidemiologia Clinica; Esperanza Martínez-Abundis, MD, MSc, PhD, Study Director — Unidad de Investigacion Medica en Epidemiologia Clinica
Locations (1):
- Unidad de Investigacion Medica en Epidemiologia Clinica, Hospital de Especialidades, UMAE, Centro Medico Nacional de Occidente, Guadalajara, Jalisco, Mexico